CLINICAL TRIAL: NCT01609699
Title: A Baseline Controlled Study to Evaluate the Effectiveness of the UltraShape® Contour I - Y System for Non-Invasive Reduction in Abdominal Circumference
Brief Title: Effectiveness Study of the UltraShape® Contour I-Y for Non-Invasive Reduction in Abdominal Circumference
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UltraShape (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US-RB-CY1
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Reduction in Abdominal Circumference
Keywords: body circumference; Non-Invasive Reduction
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - will undergo 3 successive treatments, 1 week apart (Experimental): The Contour I - Y System is a non-invasive focused ultrasound, for body contouring purposes, designed to selectively disrupt sub-dermal fat cells at a designated focus employing focused ultrasound. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.
  Interventions: Device: Treatment with Contour I-Y system
- Group B - will undergo 3 successive treatments, 2 weeks apart (Experimental): The Contour I - Y System is a non-invasive focused ultrasound, for body contouring purposes, designed to selectively disrupt sub-dermal fat cells at a designated focus employing focused ultrasound. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.
  Interventions: Device: Treatment with Contour I-Y system

INTERVENTIONS:
Device: Treatment with Contour I-Y system — The Contour I - Y System is a non-invasive focused ultrasound, for body contouring purposes, designed to selectively disrupt sub-dermal fat cells at a designated focus employing focused ultrasound. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.
  Other Names: UltraShape® Contour I - Y System
Device: Treatment with Contour I-Y system — The Contour I - Y System is a non-invasive focused ultrasound, for body contouring purposes, designed to selectively disrupt sub-dermal fat cells at a designated focus employing focused ultrasound. All other types of tissue, such as blood vessels, muscles and peripheral nerves remain intact. There are no thermal effects. Fat cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.
  Other Names: UltraShape® Contour I - Y System
  Arms: Group B - will undergo 3 successive treatments, 2 weeks apart

SUMMARY:
The UltraShape® Contour I- Y system uses focused ultrasound to produce localized mechanical motion within fat tissues and cells for the purpose of producing mechanical cellular membrane disruption. It is intended for reduction in body circumference.

The primary objective of this study is to evaluate the efficacy of the Contour I - Y System on abdominal circumference reduction relative to baseline pretreatment values using different treatment methods.

The primary efficacy endpoint in this trial is Statistical Difference of Circumference reduction between Baseline measurement and at follow-up measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, 18-65 years of age at the time of enrollment
2. Abdominal and flank fat thickness of at least 1.5 cm prior to initial treatment (measurement by caliper)
3. For women of child-bearing potential: negative pregnancy test in the 24 hour period prior to enrollment (measured in urine)
4. General good health confirmed by medical history and skin examination of the treated area
5. Written informed consent to participate in the study
6. Ability to comply with the requirements of the study
7. BMI ≤ 30

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease or malignancy
3. Previous liposuction in the treatment areas
4. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
5. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
6. Poor skin quality (i.e., laxity)
7. Abdominal wall diastasis or hernia on physical examination
8. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
9. Obesity (BMI > 30)
10. Childbirth within the last 12 months or women who suckling a child
11. Any acute or chronic condition which, in the opinion of the Investigator, could interfere with the conduct of the study
12. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
13. Inability to comply with circumference measurement procedure (e.g., inability to held breath for the required duration)
14. Participation in another clinical study
15. Previous body contouring treatments in the abdomen or love handle areas

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of the Contour I - Y System on abdominal circumference reduction relative to baseline pretreatment values using different treatment methods. | 3.5 months

SECONDARY OUTCOMES:
The secondary objective of this study subject satisfaction measured with a self-assessment questionnaire | 3.5 months
Rate of device and procedure related adverse event adverse | 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ad-El, MD, Principal Investigator — Rabin Medical Center - Beilinson Hospital
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel